CLINICAL TRIAL: NCT00188188
Title: Endothelial Dysfunction in Systemic Lupus Erythematosus: Its Contribution to Abnormalities in Coronary Perfusion.
Brief Title: Study of Endothelial Dysfunction in Systemic Lupus and Its Role in Heart Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SLED
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-12-29 (Estimated); Status verified 2005-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Endothelial; Dysfunction; Systemic; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

INTERVENTIONS:
Drug: quinipril

SUMMARY:
Systemic Lupus Erythematosus is a relatively common autoimmune disease that affects mainly women.Cardiovascular disease as a result of accelerated atherosclerosis is a major cause of mortality and morbidity in SLE.Previous research has shown that 35-40% of patients with SLE have abnormalities of myocardial perfusion even when they have no coronary stenoses on coronary angiography. The reason for these frequent perfusion abnormalities in the absence of angiographically significant CAD remains uncertain, but could conceivably result from endothelial dysfunction. In SLE, coronary endothelial dysfunction could result from the inflammatory process involved in the SLE disease itself, a finding that could explain the correlation between disease activity and the development of CAD in these patients.As such endothelial dysfunction may account for accelerated atherosclerosis and cardiac perfusion defects (without angiographically significant coronary lesions). We propose to first evaluate whether endothelial dysfunction occurs in these patients and is more frequent in patients with myocardial perfusion abnormalities. Endothelial function will be assessed by measuring flow-mediated brachial artery dilatation. In the 250 patients included in the study we will correlate endothelial function and myocardial perfusion abnormalities to SLE disease activity, to its treatment and to the presence of CAD risk factors In a subgroup of patients (estimated 5 patients) in whom it is clinically indicated, coronary angiography will be performed in order to assess the presence of significant coronary stenoses (>50%),coronary artery reserve and coronary endothelial dysfunction. We will then attempt to reverse abnormalities in endothelial function and myocardial perfusion by therapy with an ACE inhibitor(Quinapril).Patients with myocardial perfusion abnormalities will be randomised to receive Medication A(oral Quinapril or Placebo) for 8 weeks, will have all baseline investigations repeated and then will switch over and receive medication B(Quinapril or placebo) for a further 8 weeks followed by repeat investigations.

ELIGIBILITY:
Inclusion Criteria:

>20 years Lupus according to ACR criteria Patients who demonstrate abnormality on mycardial perfusion imaging are eligible for treatment arm of study

-

Exclusion Criteria:

Steroid dependent asthma known contraindication to dipyridamole known intolerance to or contraindication to use of ACE inhibitors history of angioedema serum creatinine. 200mmol/l Renal artery stenosis pregnant or breast feeding inability to perform low grade exercise presently taking ACE, ARB or nitrates

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Iwanochko, MD, Study Director — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto Western Division, Toronto, Ontario, Canada